CLINICAL TRIAL: NCT02270645
Title: Randomized Pilot Study of Treatment for Basal Cell Carcinoma Using the Multiplex 595/1064 nm Laser
Brief Title: Randomized Pilot Study of Treatment for BCC Using the Multiplex 595/1064 nm Laser
Acronym: BCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Keyvan Nouri, MD, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120815
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Nodular Basal Cell Carcinoma; Superficial Basal Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment: 595/1064 multiplex laser (Experimental): Subjects in the treatment arm will receive 3 treatments using the 595/1064 multiplex laser spaced by a four week interval (+/- 3 days), administered in an outpatient clinic setting. If a subject in the treatment arm has multiple BCCs satisfying inclusion criteria, all BCCs will be treated.
  Four weeks (+/- 3 days) after the last treatment (Day 84) both treatment and control patients will be assessed for final clinical appearance, measurement, and evaluation of the lesion by a dermatologist.
  Subjects will also undergo deep excisional biopsy encompassing the entire lesion to determine residual tumor cell presence. If histologic examination of the tissue reveals residual BCC, then the subject will receive standard of treatment.
  Interventions: Device: 595/1064 multiplex laser
- Control (No Intervention): Subjects in the control arm will receive 3 regular study visits spaced 4 weeks (+/- 3 days) apart. If a subject in the control arm has multiple BCCs satisfying inclusion criteria, all BCCs will not be treated.
  Four weeks (+/- 3 days) after the last (Day 84) both treatment and control patients will be assessed for final clinical appearance, measurement, and evaluation of the lesion by a dermatologist.
  Subjects will also undergo deep excisional biopsy encompassing the entire lesion to determine residual tumor cell presence. If histologic examination of the tissue reveals residual BCC, then the subject will receive standard of treatment.

INTERVENTIONS:
Device: 595/1064 multiplex laser — 595/1064 multiplex laser will be used 3 times spaced by a four week interval (+/- 3 days), it will be administered in an outpatient clinic setting.
  Arms: Treatment: 595/1064 multiplex laser

SUMMARY:
Laser therapy for basal cell carcinoma may be a superior option for patients who do not wish to or cannot tolerate other treatment modalities such as topical chemotherapeutics or surgery.

In this pilot study, we will preliminarily assess the efficacy and safety of the 595/1064 nm Multiplex laser when treating superficial and nodular basal cell carcinomas less than 1.5 cm in size. This is an unblinded study in which patients will be randomized to either a treatment arm or a control arm. Patients in the treatment arm will receive three treatments with the 595/1064 nm multiplex laser spaced four weeks apart. The control group will visit the clinic with the same schedule as the treatment group for monitoring of the lesion. All patients will return one month after last treatment session or clinical visit, for evaluation of clinical and histological clearance.

DETAILED DESCRIPTION:
Basal cell carcinoma is a malignancy with significant prevalence that rarely metastasizes but can be locally destructive. Laser therapy for this type of lesion may be a superior option for patients who do not wish to or cannot tolerate other modalities such as topical chemotherapeutics or surgery.

In this pilot study, we will preliminarily assess the efficacy and safety of the 595/1064 nm Multiplex laser when treating superficial and nodular basal cell carcinomas less than 1.5 cm in size. Eligible patients with biopsy-proven superficial or nodular BCCs less than 1.5 cm in size will have the opportunity to enroll in this study. This is an unblinded study in which patients will be randomized to either a treatment arm or a control arm. Patients in the treatment arm will receive three treatments with the 595/1064 nm multiplex laser spaced four weeks apart. In addition to assessing the presence of any adverse effects, photographs will be taken at each visit. One month after the last treatment session, patients in this group will return for evaluation of 1) clinical clearance and 2) histological clearance of their BCC. In order to assess clinical clearance, a dermatologist will grossly examine, measure, and document any residual lesion. Afterwards, a deep excisional biopsy encompassing the entire region will be taken and histological clearance will be determined by a microscopic examination for any residual tumor cells. Follow-up for wound care of the biopsy will occur one week later. Tumor burden will be calculated by change in surface area of the lesion.

After standard diagnostic biopsy, patients in the control arm will be followed for three regular visits, spaced 4 weeks apart. One month after the third follow-up visit, control patients will return for final photography and evaluation of clinical and histological clearance, just as the treatment arm. Although extremely rare1, if any clinical signs of progression are visible during this period (what we will consider greater than 10% growth), the patient will be withdrawn from the study and will undergo standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Diagnostic biopsy must be no later than three months prior to enrollment
* Lesion is biopsy-proven nodular or superficial BCC
* BCC is 1.5 cm or less in diameter
* BCC is on trunk or extremities
* Fitzpatrick skin types I, II, III, or IV
* If female, must no longer be of child-bearing potential
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* BCC is greater than 1.5 cm in size
* If location of BCC is on the face.
* Patients whose biopsy shows a subtype other than superficial or nodular, or has characteristics of a more aggressive nature, such as: Basosquamous basal cell carcinoma, Morpheaform/ infiltrative basal cell carcinoma, Sclerosing basal cell carcinoma, Recurrent basal cell carcinomas
* Patients who may not be able to tolerate light therapy, such as: Patients with seizure disorders triggered by light, Patients who have or are currently receiving gold therapy, Patients with any light sensitive disorder, Patients taking medication that increases sensitivity to light, Patients with Systemic Lupus Erythematous
* Fitzpatrick skin types V or VI
* Patients who are taking certain oral medications such as: Anticoagulants except for aspirin 81 mg, Isotretinoin (currently or within last 6 months), Medications that alter wound healing
* Patients who have a history of Herpes Simplex Virus outbreak in the area to be treated
* Patients whose lesion has been previously, or is currently being, treated by another modality (topical immunomodulators/ chemotherapeutics, cryotherapy, curettage and electrodesiccation, surgical excision, or Mohs micrographic surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Nouri, MD, Principal Investigator — University of Miami Silvester Comprenhensive Care Center
Locations (1):
- University of Miami Hospital and Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Lesion
Groups:
- Treatment: 595/1064 Multiplex Laser: Subjects in the treatment arm will receive 3 treatments using the 595/1064 multiplex laser spaced by a four week interval (+/- 3 days), administered in an outpatient clinic setting. If a subject in the treatment arm has multiple BCCs satisfying inclusion criteria, all BCCs will be treated.
  Four weeks (+/- 3 days) after the last treatment (Day 84) both treatment and control patients will be assessed for final clinical appearance, measurement, and evaluation of the lesion by a dermatologist.
  Subjects will also undergo deep excisional biopsy encompassing the entire lesion to determine residual tumor cell presence. If histologic examination of the tissue reveals residual BCC, then the subject will receive standard of treatment.
  595/1064 multiplex laser: 595/1064 multiplex laser will be used 3 times spaced by a four week interval (+/- 3 days), it will be administered in an outpatient clinic setting.
Period: Overall Study
Arm/Group | Treatment: 595/1064 Multiplex Laser | Control
Started | 8; 11 Lesion | 4; 5 Lesion
Completed | 6; 9 Lesion | 4; 5 Lesion
Not Completed | 2; 2 Lesion | 0; 0 Lesion

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment: 595/1064 Multiplex Laser | Control | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 57.7 [32 to 76] | 63.5 [60 to 69] | 59.6 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Lesions Cleared Histologically
Description: Number of lesions cleared clinically and histologically. The lesion clearance was determined by measuring the size of lesion which also included a histological evaluation 4 weeks after the treatment.
Time Frame: 91 days
Population: In the treatment arm, there were 6 patients with a total of 9 lesions. Some of these patients had multiple lesions treated.
  In the control arm, there were 4 patients with a total of 5 lesions. Some of these patients had multiple lesions treated.
Measure: Count of Units; unit: Lesion
Units Other Than Participants: Lesion
Arm/Group | Treatment: 595/1064 Multiplex Laser | Control
Number analyzed (Participants) | 6 | 4
Number analyzed (Lesion) | 9 | 5
Lesion | 3 | 5

2. Secondary Outcome: Number of Adverse Events Reported
Description: Adverse events reported by participants
Time Frame: 91 days
Measure: Number; unit: Adverse Events
Arm/Group | Treatment: 595/1064 Multiplex Laser | Control
Number analyzed (Participants) | 8 | 4
Adverse Events | 1 | 0

ADVERSE EVENTS:
Time Frame: 91 days
Arm/Group | Treatment: 595/1064 Multiplex Laser | Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 1/8 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: 595/1064 Multiplex Laser (N=8) | Control (N=4)
Fibrosing on histology result (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT02270645/Prot_SAP_000.pdf